CLINICAL TRIAL: NCT04527718
Title: A Phase 1 Randomized, Double Blinded, Placebo-Controlled Single Dose Escalation Study to Evaluate the Safety, Tolerability and Pharmacokinetic Characteristics of 611 in Adult Healthy Male and Female Volunteers
Brief Title: Study of the Safety, Tolerability and Pharmacokinetics of 611 in Adult Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sunshine Guojian Pharmaceutical (Shanghai) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SSGJ-611-HV-I-A
Record Dates: First submitted 2020-07-16; First posted 2020-08-26 (Actual); Last update posted 2022-11-10 (Actual); Status verified 2022-11

CONDITIONS: Healthy
MeSH Terms: interventions — entacapone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Cohort 1 (Experimental): 611 dose 1 (45mg) plus placebo
  Interventions: Drug: Placebo; Drug: 611
- Cohort 2 (Experimental): 611 dose 2 (150mg) plus placebo
  Interventions: Drug: Placebo; Drug: 611
- Cohort 3 (Experimental): 611 dose 3 (300mg) plus placebo
  Interventions: Drug: Placebo; Drug: 611
- Cohort 4 (Experimental): 611 dose 4 (450mg) plus placebo
  Interventions: Drug: Placebo; Drug: 611
- Cohort 5 (Experimental): 611 dose 5 (600mg) plus placebo
  Interventions: Drug: Placebo; Drug: 611

INTERVENTIONS:
Drug: Placebo — placebo as a single SC injection on Day 1;
Drug: 611 — 611 as a single SC injection on Day 1;

SUMMARY:
This is a Phase 1 randomized, double blinded, placebo-controlled, single dose escalation study to evaluate the safety, tolerability, and PK of 611 in healthy volunteers.

DETAILED DESCRIPTION:
Total duration of the study period per subject is about 4 months broken down as follows:

The screening period is up to 28 days, one dose treatment, and follow- up period is up to 71±7 days (90±9 days for Cohorts 1 and 2).

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand and willing to sign the ICF
2. Healthy male and female subjects, non-smokers, 18-55 years of age
3. In the opinion of the investigator, with no significant medical history, and in good health.
4. Body mass index 19.0-32.0 kg/m2 and body weight ≥ 50.0 kg for males and ≥ 45.0 kg for females.
5. Subjects are able to follow the study protocol and complete the trial.

Exclusion Criteria:

1. History of hypersensitivity to similar drugs to 611 or their excipients.
2. Pregnant, or nursing females.
3. HepBsAg or HepCAb positive.
4. Human immunodeficiency virus (HIV) positive.
5. Positive urine drug screen, or cotinine test.
6. Any reason which, in the opinion of the Qualified Investigator, would prevent the subject from participating in the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2020-09-09 (Actual); Primary Completion 2021-08-13 (Actual); Study Completion 2021-08-13 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With TEAEs | up to 71days (90 days for Cohorts 1 and 2)
  Incidence of treatment-emergent adverse events (TEAEs) will be summarized by SOC and PT for each treatment group, and also be summarized by severity and association with the study treatments.

SECONDARY OUTCOMES:
PK | up to 71days (90 days for Cohorts 1 and 2)
  PK parameters not limit to Cmax
Incidence of immunogenicity | up to 71days (90 days for Cohorts 1 and 2)
  ADA, and NAbs if ADA is positive

CONTACTS AND LOCATIONS:
Locations (1):
- Covance Dallas Clinical Research Unit, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No